CLINICAL TRIAL: NCT05820334
Title: Fatigue in Multiple Sclerosis Patients; Subjective, Objective and Cognitive Analysis
Brief Title: Multiple Sclerosis and Fatigue Assessment
Status: Completed | Type: Observational
Sponsor: Asli Demirtaş (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Asli Demirtaş, Lecturer, MSc., PT., Nigde Omer Halisdemir University
Organization: Nigde Omer Halisdemir University (Other)
Other Study IDs: Gazi University (2023-157)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Fatigue; Assessment; Objective; Cognitive
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fatigue in patients with Multiple Sclerosis (MS) is a problem that is seen without physical exertion and affects the majority of patients. In studies on fatigue in the literature, it has been seen that subjective methods are frequently used by using evaluation scales based on patient statements, but objective evaluation methods are not yet sufficient. This study was planned to compare the measurement results by evaluating fatigue subjectively, objectively and cognitively in MS patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, inflammatory, demyelinating, autoimmune disease of the central nervous system. It is characterized by clinical symptoms arising from lesions in the brain, spinal cord or optic nerves. Although fatigue is one of the most common and most disabling problems of individuals with MS, it is not yet fully understood. This affects the treatment and disease process in MS. Despite studies to elucidate the pathogenic mechanisms of fatigue, available information is limited. Several factors contribute to the limited fatigue research, but the most important is that 'fatigue' is often not clearly defined or meaningful measures cannot be made in clinical/research settings. The first step in the evaluation of fatigue, which is a complex symptom, is to start with the identification and analysis of the factors that may cause fatigue, and to comprehensively question the factors that may be effective and the patient's history, and to evaluate the fatigue subjectively and objectively after the comprehensive patient history. The fatigue of patients diagnosed with MS will be evaluated subjectively, objectively and cognitively. Other information about the disease of the patients will be recorded. Subjective fatigue assessment methods, objective fatigue assessment methods and cognitive fatigue assessment methods will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having a definite diagnosis of Relapsing Remitting MS by a neurologist,
* Expanded Disability Status Scale (EDSS) score between 1-5.5,
* To be stable in medical treatment,
* Being able to stand independently for at least 60 seconds without any assistive device,
* It is to be above 24 points according to the Mini-Mental State Examination (MMSE) evaluation.

Exclusion Criteria:

* Being diagnosed with MS for less than 1 year,
* Having had an MS attack in the last 3 months,
* Being illiterate or unable to communicate in Turkish,
* Having an active infection,
* Being pregnant,
* Having an orthopedic problem or having a surgery that may affect the lower extremity,
* Having an additional neurological or circulatory disease that may cause balance disorder, a problem affecting the vision or vestibular tract, or a diagnosis of orthopedic surgery, rheumatological disease,
* To be included in the physiotherapy and rehabilitation program in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients who applied to Nigde Omer Halisdemir University Training and Research Hospital Neurology Clinic or Hacettepe University Faculty of Medicine Neurology Department or who are referred to Gazi University Department of Physiotherapy and Rehabilitation will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity | Baseline
  In the Fatigue Severity Scale (FSS), participants are asked to rate their fatigue level between 1 and 7 in the 9 statements (including motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life) during the last week.The minimum score possible is 9 and the highest is 63. The higher score indicates more severe fatigue.
Fatigue Impact | Baseline
  The Fatigue Impact Scale (FIS) was first developed by Fisk to evaluate the symptoms of fatigue in disease states and the effects of fatigue on daily life. FIS considers the fatigue in the last month. It consists of 40 questions in total, investigating the effects of fatigue on cognitive (10 questions), physical (10 questions), and psychosocial (20 questions). Since each question is scored between 0 (no problem) and 4 (maximum problem), the total score of the scale is 160, and an increase in the score means that the effect of fatigue increases. Cognitive function, memory, thinking and regulation; physical function motivation, endurance and effort; psychosocial function evaluates the effect of fatigue on emotions, coping and workload based on self-report.
Fatigue Assessment | Baseline
  "Checklist Individual Strength" (CIS) Scale: It was developed by Beurskens and adapted into Turkish by Ergin to measure the general fatigue levels of individuals. It is a valid and reliable fatigue assessment scale in patients with MS. According to this scale, fatigue; subjective perception of fatigue is evaluated in four aspects as decrease in concentration, decrease in motivation and decrease in physical activity. The questionnaire consists of 20 statements measuring the fatigue in the last 2 weeks and a 7-point scale is used for the answers. The lowest score that can be obtained from the scale is 20, and the highest score is 140.
Cognitive Fatigue Assessment | Baseline
  The Brief International Cognitive Assessment for MS (BICAMS) initiative was undertaken to recommend a brief, cognitive assessment for MS that is optimized for small centers. BICAMS was particularly focused on international use, to facilitate comparison across settings. An expert committee of twelve neurologists and neuropsychologists representing the main cultural groups that have so far contributed extensive data about cognitive dysfunction in MS was convened. The opinions generated from the meeting are published elsewhere. Consensus was also achieved on optimal measures for learning and memory in MS patients, time permitting: the initial learning trials of the second edition of the California Verbal Learning Test (CVLT2) and the revised Brief Visuospatial Memory Test (BVMTR).
Lower extremity functions | Baseline
  The 25-Step Walking Test is a test that measures lower extremity functions. It has been developed for the purpose of recording the patient with this test at each examination. The patient is asked to walk in a predetermined interval. The average of both times is taken by noting the number of seconds spent on the way out and on the way back.
Upper extremity functions | Baseline
  Upper extremity function was evaluated with the 9-Hole Peg Test (9-HPT). It consists of moving nine pegs into one of the nine holes on a peg board, then back into an open box. A stopwatch was used for the measurements and the scores were recorded in seconds (s).
Hand grip-fatigue assessment | Baseline
  In order to evaluate the fatigue that may occur due to time, the grip muscle strength that individuals can sustain for a certain period of time will be evaluated. A 'K-Force Grip grip dynamometer' will be used for the measurement. The values and fatigue level will be recorded by making three attempts for both hands in the determined position. The test will be administered for 30 seconds. A 1-minute rest will be given between measurements. The average value for fatigue and grip strength will be calculated.
Muscle strength-fatigue assessment | Baseline
  Fatigue is automatically calculated and reported by the K-Force device. The device software fatigue value is calculated based on the changes in performance during muscle contraction. In the evaluation of muscle strength, the 'K-Force Muscle Controller' will be evaluated using a muscle dynamometer. For the lower extremity, hip flexion, hip abduction, and knee extension will be evaluated bilaterally. Shoulder flexion, shoulder abduction and elbow flexion muscle strength will be evaluated for the upper extremity. In the lower and upper extremities, the measurement will be repeated 3 times for both sides and the average value will be calculated and recorded. A 1-minute rest will be given between measurements. The fatigue value determined for each measurement will also be recorded. Test positions applied during manual muscle testing will be applied to provide standardization for assessment.
Balance-fatigue assessment | Baseline
  In order to evaluate the fatigue that may occur due to performance, the balance of individuals and the resulting fatigue will be evaluated using the Visual Analog Scale-Fatigue (VAS-F) before and after the balance changes calculated from the device during the balance tests. It will be evaluated using the 'Force Plates' device in the evaluation of balance. Foot sole pressure distributions, ground reaction forces, static and dynamic balance evaluations, symmetry will be evaluated. For static balance; balance on one leg, balance on both legs with eyes open and eyes closed will be evaluated. dynamic balance; will be evaluated by the squat assessment. Measurements will be repeated 3 times and the average value will be calculated and recorded. A 1-minute rest will be given between measurements. The higher scores mean a worse in assessment.

SECONDARY OUTCOMES:
Extended Disability Status Scale (EDSS) | Baseline
  Expanded Disability Status Scale (EDSS) is the most commonly used scale to monitor disease stage and assess disability in multiple sclerosis patients. Eight functional systems (FS) are evaluated with EDSS (Visual functions, brain stem functions, pyramidal functions, cerebellar functions, sensory functions, bladder and bowel functions, cerebral functions and other). In addition, gait is also evaluated and a score between 0 (normal neurological status) and 10 (death due to MS) is determined by considering functional system scores and the level of independence of the patient in ambulation.
Standardized Mini Mental Test | Baseline
  There are 19 items in this test, which consists of 5 main parts: orientation, recording memory, attention and calculation, recall and language. The total score of the test is evaluated out of 30 and 24 points are accepted as the threshold value for the diagnosis of mild dementia. The higher the score, the higher the cognition of individuals.
Subjective fatigue assessment | Baseline
  A visual analog scale will be used.Their values range from 0-10. The higher scores mean a worse in assessment.

OTHER OUTCOMES:
Interview form | Baseline
  With a questionnaire prepared by the researchers and applied by face-to-face interview method; age (year), height (cm), body weight (kg), body mass index (BMI- kg/m2), year of diagnosis, frequency of attacks, date of last attack, marital status (married/single), education level Information such as (literate, primary school, secondary school, high school, associate degree, undergraduate, graduate), dominant extremity (right, left), CV and family history, use of assistive devices, smoking and alcohol habits, drugs used, and surgeries will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: İlke KESER, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No